CLINICAL TRIAL: NCT03599518
Title: A Multicenter, Open-Label Phase 1 Study of DS-1205c in Combination With Gefitinib in Subjects With Metastatic or Unresectable EGFR-Mutant Non-Small Cell Lung Cancer
Brief Title: DS-1205c With Gefitinib for Metastatic or Unresectable Epidermal Growth Factor Receptor (EGFR)-Mutant Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated based on a business decision by the Sponsor.
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS1205-A-J102; 184026 (Registry Identifier: JAPIC CTI)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-1205c with Gefitinib (Experimental): Participants receive DS-1205c (at planned doses given orally twice daily: 200 mg, 400 mg, 800 mg, 1000 mg, 1200 mg) in combination with daily 250 mg oral dose of gefitinib
  Interventions: Drug: DS-1205c; Drug: Gefitinib

INTERVENTIONS:
Drug: DS-1205c — DS-1205c 200 mg capsule for oral administration
  Other Names: Experimental product
Drug: Gefitinib — Gefitinib 250 mg tablet for oral administration

SUMMARY:
This study has two parts: dose escalation and dose expansion.

The primary objectives are:

* For Dose Escalation, to assess the safety and tolerability of DS-1205c when combined with gefitinib in the study population and to determine the recommended dose for expansion of DS-1205c when combined with gefitinib in the study population
* For Dose Expansion, to assess the safety and tolerability of DS-1205c when combined with gefitinib in the study population.

In Dose Escalation, after a 7-day run in period (Cycle 0), there will be 21-day cycles (Cycle 1 onward). In Dose Expansion, there will be 21-day cycles.

The number of treatment cycles is not fixed in this study. Participants will continue study treatment for 36 months unless they decide not to (withdraw consent), their disease gets worse [progressive disease (PD)], or side effects become unacceptable (unacceptable toxicity).

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically documented adenocarcinoma NSCLC
2. Has locally advanced or metastatic NSCLC, not amenable to curative surgery or radiation
3. Has acquired resistance to EGFR tyrosine kinase inhibitor (TKI) according to the Jackman criteria (PMID: 19949011):

   1. Historical confirmation that the tumor harbors an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q) OR
   2. Has experienced clinical benefit from an EGFR TKI, followed by systemic progression [Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) or World Health Organization (WHO)] while on continuous treatment with an EGFR TKI
4. Is currently receiving and able to interrupt gefitinib or discontinue erlotinib, afatinib, or osimertinib
5. Has been receiving gefitinib, erlotinib, afatinib, or osimertinib for at least 6 weeks with well-controlled related toxicities less than Grade 3 in severity at the time of screening period; participants who have been receiving gefitinib must be taking gefitinib at a dose of 250 mg/day
6. Has radiological documentation of disease progression while receiving continuous treatment with gefitinib, erlotinib, afatinib, or osimertinib
7. Has at least one measurable lesion per RECIST version 1.1
8. Is willing to provide archival tumor tissue from a biopsy performed after progression during treatment with gefitinib, erlotinib, afatinib, or osimertinib OR has at least one lesion, not previously irradiated, amenable to core biopsy and is willing to undergo screening tumor biopsy
9. Demonstrates absence of EGFR T790M mutation in tumor tissue since progression during gefitinib, erlotinib, afatinib, or osimertinib treatment
10. Has Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1, with no deterioration over the previous 2 weeks

Exclusion Criteria:

1. Has any evidence of small cell histology, or combined small cell and non-small cell histology, in original tumor biopsy or in screening biopsy performed since progression
2. Has previously documented evidence of anaplastic lymphoma kinase (ALK) fusion, ROS proto-oncogene 1 (ROS1) fusion, BRAF V600E mutation, rearranged during transfection (RET) rearrangement, human epidermal growth factor receptor 2 (HER2) mutation, or MET exon 14 skipping mutation - no new testing for these genomic alterations is required for Screening
3. Has received treatment with any of the following:

   1. Any cytotoxic chemotherapy, immune checkpoint inhibitor therapy, investigational agent or other anticancer drug(s) from a previous cancer treatment regimen or clinical study (other than EGFR TKI), within 14 days of the first dose of study treatment
   2. Immune checkpoint inhibitor therapy within 30 days of first dose of study treatment
   3. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
   4. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks, or palliative radiation therapy within 2 weeks of the first dose of study drug treatment
4. Has history of other active malignancy within 3 years prior to enrollment, except:

   1. Adequately treated non-melanoma skin cancer OR
   2. Superficial bladder tumors (Tumor stage "a" [Ta], Tumor stage "is" [Tis], Tumor stage "1" [T1]) OR
   3. Curatively treated in situ disease OR
   4. Low-risk non-metastatic prostate cancer (with Gleason score < 7 on antiandrogen therapy)
5. Has spinal cord compression or clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms - Subjects with clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (1 week for stereotactic radiotherapy).
6. Has retinal disease in the eye that is not due to neovascular age-related macular degeneration (nAMD; eg, significant diabetic retinopathy, glaucomatous retinal atrophy, retinal detachment)
7. Has history of myocardial infarction within the past 6 months
8. Has symptomatic congestive heart failure [New York Heart Association (NYHA) Classes II-IV], unstable angina, or cardiac arrhythmia requiring antiarrhythmic treatment
9. Has left ventricular ejection fraction (LVEF) < 45% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan
10. Has any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, eg, complete left bundle branch block, third-degree heart block, second-degree heart block, or PR interval > 250 milliseconds (ms)
11. Has a mean corrected QT interval using Fridericia's correction (QTcF) prolongation >470 ms for females and >450 ms for males in three successive Screening measurements
12. Unable or unwilling to discontinue concomitant use of drugs that are known to prolong the QT interval
13. Has any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as congenital long QT. syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives
14. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroid treatment, has current ILD/pneumonitis, or has suspected ILD/pneumonitis which cannot be ruled out by imaging at screening
15. Has history of pancreatitis within the past 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (8):
- Japan (8):
  - Aichi Cancer Center, Chikusa, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kindai University Hospital, Sayama, Osaka
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Ariake, Tokyo
  - National Cancer Center Hospital, Tsukiji, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Shizuoka Cancer Center, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Goto K, Shiraishi Y, Murakami H, Horinouchi H, Toyozawa R, Takeda M, Uno M, Crawford N, McGill J, Jimbo T, Ishigami M, Takayama G, Nakayama S, Ohwada S, Nishio M. Phase 1 study of DS-1205c combined with gefitinib for EGFR mutation-positive non-small cell lung cancer. Cancer Med. 2023 Mar;12(6):7090-7104. doi: 10.1002/cam4.5508. Epub 2023 Jan 9. PMID 36621830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants were enrolled and treated in this clinical trial from 21 Sep 2018 to 29 Jun 2020 at 8 clinic sites in Japan.
Pre-assignment Details: Dose Escalation started with a DS-1205c monotherapy 7-day run-in period (Cycle 0), followed by combination treatment (DS-1205c + gefitinib). Participants received a final dose of gefitinib, erlotinib, afatinib, dacomitinib, or osimertinib on Cycle 0, Day -1. During the run-in period, participants received DS-1205c orally twice daily (BID). On Cycle 1, Day 1, DS-1205c was administered orally BID in combination with gefitinib 250 mg administered orally once daily (21-day cycles).
Groups:
- DS-1205c 200 mg + Gefitinib: Participants who received DS-1205c 200 mg twice daily (BID) in combination with daily 250 mg oral dose of gefitinib.
- DS-1205c 400 mg + Gefitinib: Participants who received DS-1205c 400 mg twice daily (BID) in combination with daily 250 mg oral dose of gefitinib.
- DS-1205c 800 mg + Gefitinib: Participants who received DS-1205c 800 mg twice daily (BID) in combination with daily 250 mg oral dose of gefitinib.
- DS-1205c 1000 mg + Gefitinib: Participants who received DS-1205c 1000 mg twice daily (BID) in combination with daily 250 mg oral dose of gefitinib.
- DS-1205c 1200 mg + Gefitinib: Participants who received DS-1205c 1200 mg twice daily (BID) in combination with daily 250 mg oral dose of gefitinib.
Period: Overall Study
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Started | 5 | 4 | 6 | 1 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 6 | 1 | 4
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease as per RECIST v1.1 | 5 | 4 | 5 | 1 | 2
Not completed — Participant withdrawal from study treatment | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib | Total
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 4 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 1 | 2 | 6
  >=65 years | 3 | 4 | 5 | 0 | 2 | 14
Age, Continuous [Median (Full Range); unit: years] | 67 [60 to 74] | 69.5 [67 to 82] | 70 [36 to 75] | 41 [41 to 41] | 66 [52 to 81] | 68.5 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 1 | 3 | 16
  Male | 2 | 0 | 1 | 0 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 6 | 1 | 4 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 5 | 4 | 6 | 1 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) Following Administration With DS-1205c in Combination With Gefitinib
Description: A dose-limiting toxicity (DLT) was defined as any treatment-emergent adverse event (TEAE) not attributable to disease or disease-related processes that occurs during the DLT-evaluation period (Cycle 0 Day 1 to Cycle 1 Day 21 of Dose Escalation) and is Grade 3 or above, according to NCI-CTCAE version 5.0.
Time Frame: Cycle 0 Day 1 (7-day cycle) to Cycle 1 Day 21 (each cycle is 21 days)
Population: Dose-limiting toxicities (DLTs) were assessed in the DLT-Evaluable Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 4 | 4 | 6 | 1 | 4
Participants | 0 | 0 | 1 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events Occurring in Participants Following Administration With DS-1205c in Combination With Gefitinib
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A treatment-emergent adverse event (TEAE) was defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity after the initiating the study drug until 37 days after last dose of the study drug.
Time Frame: Screening, Cycle 0 (7-day cycle), Days -1, 1, 2, 4, 6, and 7; Cycle 1 (21-day cycle), Days 1, 4, 8, and 15; Cycle 2 (21-day cycle), Days 1, 2, and 8; Cycle 3 and beyond (21-day cycles), Day 1; and end-of-treatment, 30 days after last dose, up to 1 year
Population: Adverse events (AEs) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 4
Participants
  Any TEAE | 5 | 4 | 6 | 0 | 4
  Infections and Infestations | 2 | 1 | 0 | 0 | 1
  Upper respiratory tract infection | 1 | 0 | 0 | 0 | 1
  Nasopharyngitis | 0 | 1 | 0 | 0 | 0
  Paronychia | 1 | 0 | 0 | 0 | 0
  Neoplasms Benign, Malignant, and Unspecified (including Cysts and Polyps) | 1 | 1 | 1 | 0 | 0
  Tumour pain | 1 | 1 | 1 | 0 | 0
  Blood and Lymphatic System Disorders | 0 | 0 | 1 | 0 | 1
  Anaemia | 0 | 0 | 0 | 0 | 1
  Neutropenia | 0 | 0 | 1 | 0 | 0
  Metabolism and Nutrition Disorders | 3 | 0 | 0 | 0 | 0
  Decreased appetite | 1 | 0 | 0 | 0 | 0
  Hypertriglyceridaemia | 1 | 0 | 0 | 0 | 0
  Hyperuricaemia | 1 | 0 | 0 | 0 | 0
  Nervous System Disorders | 2 | 0 | 0 | 0 | 0
  Hypoaesthesia | 1 | 0 | 0 | 0 | 0
  Vagus nerve disorder | 1 | 0 | 0 | 0 | 0
  Eye Disorders | 0 | 2 | 1 | 0 | 0
  Conjunctival haemorrhage | 0 | 1 | 0 | 0 | 0
  Dry eye | 0 | 1 | 0 | 0 | 0
  Eye disorder | 0 | 0 | 1 | 0 | 0
  Ear and Labyrinth Disorders | 1 | 0 | 0 | 0 | 0
  Vertigo | 1 | 0 | 0 | 0 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 0 | 1 | 0 | 0 | 0
  Cough | 0 | 1 | 0 | 0 | 0
  Gastrointestinal Disorders | 4 | 3 | 3 | 0 | 3
  Diarrhoea | 0 | 3 | 1 | 0 | 1
  Nausea | 1 | 0 | 0 | 0 | 2
  Vomiting | 2 | 0 | 1 | 0 | 0
  Constipation | 2 | 0 | 0 | 0 | 0
  Dyspepsia | 1 | 0 | 0 | 0 | 1
  Stomatitis | 1 | 1 | 0 | 0 | 0
  Abdominal pain lower | 0 | 0 | 1 | 0 | 0
  Abdominal pain upper | 0 | 0 | 0 | 0 | 1
  Hepatobiliary Disorders | 0 | 0 | 0 | 0 | 1
  Hepatic function abnormal | 0 | 0 | 0 | 0 | 1
  Skin and Subcutaneous Tissue Disorders | 3 | 3 | 5 | 0 | 3
  Rash maculo-papular | 1 | 0 | 3 | 0 | 2
  Dermatitis acneiform | 0 | 3 | 0 | 0 | 0
  Pruritus | 1 | 0 | 1 | 0 | 0
  Rash | 0 | 0 | 1 | 0 | 1
  Dry skin | 0 | 1 | 0 | 0 | 0
  Skin hyperpigmentation | 1 | 0 | 0 | 0 | 0
  Musculoskeletal and Connective Tissue Disorders | 0 | 1 | 0 | 0 | 0
  Neck pain | 0 | 1 | 0 | 0 | 0
  General Disorders and Administration Site Conditions | 1 | 0 | 2 | 0 | 1
  Pyrexia | 1 | 0 | 1 | 0 | 1
  Malaise | 0 | 0 | 1 | 0 | 0
  Pain | 0 | 0 | 1 | 0 | 0
  Investigations | 3 | 2 | 4 | 0 | 2
  Aspartate aminotransferase increased | 2 | 1 | 2 | 0 | 2
  Alanine aminotransferase increased | 1 | 1 | 2 | 0 | 2
  White blood cell count decreased | 0 | 0 | 3 | 0 | 1
  Electrocardiogram QT prolonged | 0 | 0 | 2 | 0 | 0
  Neutrophil count decreased | 0 | 0 | 1 | 0 | 1
  Amylase increased | 1 | 0 | 0 | 0 | 0
  Blood alkaline phosphatase increased | 0 | 0 | 1 | 0 | 0
  Blood creatinine phosphokinase increased | 0 | 1 | 0 | 0 | 0
  Lipase increased | 0 | 0 | 1 | 0 | 0
  Weight decreased | 1 | 0 | 0 | 0 | 0
  Injury, Poisoning and Procedural Complications | 0 | 0 | 1 | 0 | 0
  Fall | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Number of Participants With Best Overall Response With Confirmation as Assessed by Investigator Following Administration of DS-1205c in Combination With Gefitinib
Description: Complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions. Objective response rate was calculated as the number of participants with best objective response (CR + PR) determined by Investigator assessment based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1].
Time Frame: Screening; Cycle 0 (7-day cycle); Cycle 1 and beyond (21-day cycles), Every 6 weeks (± 7 days) in the first 24 weeks after Day 1 of Cycle 1, and every 12 weeks (± 7 days) thereafter; and end-of-treatment, 30 days after last dose, up to 1 year
Population: Best overall response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 4
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 0 | 0
  Stable disease (SD) | 2 | 1 | 1 | 0 | 1
  Progressive disease (PD) | 3 | 3 | 5 | 1 | 2
  Non-Evaluable (NE) | 0 | 0 | 0 | 0 | 1
  Objective response rate (CR+PR) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Disease Control Rate Assessed by Investigator Following Administration of DS-1205c in Combination With Gefitinib
Description: Disease control rate (DCR) was defined number of participants with CR+PR+SD objective response. As per the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: as for outcome 3
Population: Disease control rate (DCR) was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 4
Participants | 2 | 1 | 1 | 0 | 1

5. Secondary Outcome: Progression-free Survival Assessed by Investigator Following Administration of DS-1205c in Combination With Gefitinib
Description: Progression-free survival (PFS) was defined as the time from the date of the first dose to the earlier of the dates of the first objective documentation of radiographic PD or death due to any cause. As per the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 3
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 4
weeks | 6.7 [3.4 to 12.1] | 7.1 [6.1 to 12.9] | 6.9 [2.9 to 25] | 6.7 [NA to NA] — 95% confidence interval could not be calculated due to the small sample size | 6.9 [6.1 to 6.9]

6. Secondary Outcome: Overall Survival in Participants Following Administration of DS-1205c in Combination With Gefitinib
Description: Overall Survival (OS) was defined as the time from the date of first dose to the date of death from any cause.
Time Frame: as for outcome 3
Population: Overall survival (OS) was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 5 | 4 | 6 | 1 | 4
weeks | 27.4 [16.7 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is not applicable | NA [48.4 to NA] — Due to insufficient number of events | NA [23.4 to NA] — Due to insufficient number of events | 35.4 [NA to NA] — Not enough events occurred to estimate a standard error for the median survival time | NA [NA to NA] — Due to insufficient number of events

7. Secondary Outcome: Pharmacokinetic Parameter of Maximum Concentration (Cmax) of DS-1205a Following Administration of DS-1205c in Combination With Gefitinib
Description: Blood samples for pharmacokinetic (PK) analyses of DS-1205a were obtained at specified time points. Plasma concentrations of DS-1205a were measured using validated assays and non-compartmental analysis.
Time Frame: Predose, 1, 2, 4, 6, 8, and 10 hours of Cycle 0 (7-day cycle; DS-1205c alone), Days 1 and 7; Predose of Cycle 1 (21-day cycle), Day 1 (DS-1205c + gefitinib); Predose, 1, 2, 4, 6, 8, and 10 hours of Cycle 2 (21-day cycle; DS-1205c + gefitinib), Day 1
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 4 | 4 | 6 | 1 | 4
ng/mL
  Cycle 0, Day 1 | 316 (46.1) | 500 (141) | 623 (251) | 521 (0) | 779 (280)
  Cycle 0, Day 7: number analyzed (Participants) | 3 | 4 | 4 | 1 | 4
  Cycle 0, Day 7 | 521 (17.1) | 838 (130) | 1120 (407) | 580 (0) | 1080 (268)
  Cycle 1, Day 1: number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
  Cycle 1, Day 1 | 462 (48.1) | 907 (266) | 995 (375) | 677 (0) | 1270 (99)
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 4 | 3 | 1 | 1
  Cycle 2, Day 1 | 490 (19.8) | 688 (130) | 1030 (357) | 632 (0) | 1090 (0)

8. Secondary Outcome: Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) of DS-1205a Following Administration of DS-1205c in Combination With Gefitinib
Description: as for outcome 7
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 4 | 4 | 6 | 1 | 4
hours
  Cycle 0, Day 1 | 3.99 [3.92 to 4.05] | 4.99 [3.97 to 5.93] | 3.99 [2.02 to 6.08] | 4.15 [4.15 to 4.15] | 5.08 [4.00 to 9.80]
  Cycle 0, Day 7: number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
  Cycle 0, Day 7 | 3.97 [3.88 to 4.02] | 4.02 [3.98 to 4.25] | 5.08 [4.02 to 8.00] | 4.02 [4.02 to 4.02] | 1.97 [0 to 3.93]
  Cycle 1, Day 1: number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
  Cycle 1, Day 1 | 3.90 [3.90 to 4.00] | 4.00 [3.88 to 6.00] | 4.01 [3.97 to 4.05] | 6.03 [6.03 to 6.03] | 3.08 [0 to 6.17]
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 4 | 3 | 1 | 1
  Cycle 2, Day 1 | 1.93 [0 to 3.87] | 4.99 [0 to 6.10] | 4.13 [3.98 to 6.02] | 4.02 [4.02 to 4.02] | 0 [0 to 0]

9. Secondary Outcome: Pharmacokinetic Parameter Area Under the Plasma Concentration Curve of DS-1205a Following Administration of DS-1205c in Combination With Gefitinib
Description: Blood samples for pharmacokinetic (PK) analyses of DS-1205a were obtained at specified time points. Plasma concentrations of DS-1205a were measured using validated assays and non-compartmental analysis. Area under the plasma concentration curve from time 0 to 8 hours (AUC8h), area under the plasma concentration-time curve from time 0 to 10 hours (AUC10h), and area under the plasma concentration-time curve during a dosing interval (AUCtau) were assessed.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 4 | 4 | 6 | 1 | 4
ng*h/mL
  Cycle 0, Day 1: AUC10h | 1710 (170) | 2800 (675) | 3860 (1730) | 2440 (0) | 4280 (893)
  Cycle 0, Day 7: AUC10h: number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
  Cycle 0, Day 7: AUC10h | 3760 (136) | 5990 (945) | 8120 (2520) | 4560 (0) | 8250 (1060)
  Cycle 0, Day 7: AUCtau: number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
  Cycle 0, Day 7: AUCtau | 4430 (173) | 7000 (1010) | 9490 (2860) | 5490 (0) | 10300 (1740)
  Cycle 1, Day 1: AUC8h: number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
  Cycle 1, Day 1: AUC8h | 2980 (165) | 5670 (1360) | 6820 (2590) | 4520 (0) | 8390 (340)
  Cycle 1, Day 1: AUCtau: number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
  Cycle 1, Day 1: AUCtau | 4290 (224) | 7930 (1600) | 9820 (3640) | 6770 (0) | 12800 (691)
  Cycle 2, Day 1: AUC10h: number analyzed (Participants) | 2 | 4 | 3 | 1 | 1
  Cycle 2, Day 1: AUC10h | 3780 (536) | 5290 (1230) | 7350 (2160) | 5030 (0) | 7650 (0)
  Cycle 2, Day 1: AUCtau: number analyzed (Participants) | 2 | 4 | 3 | 1 | 1
  Cycle 2, Day 1: AUCtau | 4520 (649) | 6300 (1460) | 8530 (2640) | 6060 (0) | 9800 (0)

10. Secondary Outcome: Pharmacokinetic Parameter Trough Plasma Concentration (Ctrough) of DS-1205a Following Administration of DS-1205c in Combination With Gefitinib
Description: as for outcome 7
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set in patients with available samples for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
Number analyzed (Participants) | 3 | 4 | 4 | 1 | 2
ng/mL
  Cycle 0, Day 7 | 335 (16.7) | 497 (44.2) | 691 (155) | 437 (0) | 1040 (330)
  Cycle 1, Day 1 | 315 (21.8) | 551 (61.6) | 768 (249) | 486 (0) | 1130 (293)
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 4 | 3 | 1 | 1
  Cycle 2, Day 1 | 408 (136) | 503 (92.7) | 643 (217) | 496 (0) | 1090 (0)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from Screening, Cycle 0 (7-day cycle), Days -1, 1, 2, 4, 6, and 7; Cycle 1 (21-day cycle), Days 1, 4, 8, and 15; Cycle 2 (21-day cycle), Days 1, 2, and 8; Cycle 3 and beyond (21-day cycles), Day 1; and end-of-treatment, 30 days after last dose, up to 1 year.
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A TEAE was defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity after the initiating the study drug until 37 days after last dose of the study drug
Arm/Group | DS-1205c 200 mg + Gefitinib | DS-1205c 400 mg + Gefitinib | DS-1205c 800 mg + Gefitinib | DS-1205c 1000 mg + Gefitinib | DS-1205c 1200 mg + Gefitinib
All-Cause Mortality (participants affected / at risk) | 4/5 | 1/4 | 1/6 | 1/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/6 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 6/6 | 0/1 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-1205c 200 mg + Gefitinib (N=5) | DS-1205c 400 mg + Gefitinib (N=4) | DS-1205c 800 mg + Gefitinib (N=6) | DS-1205c 1000 mg + Gefitinib (N=1) | DS-1205c 1200 mg + Gefitinib (N=4)
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Vagus nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 3 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phophatase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate the study at the end of the Dose Escalation part and the Dose Expansion part was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT03599518/Prot_SAP_000.pdf